CLINICAL TRIAL: NCT07290218
Title: Tridimensional Robotic Assessment of Neglect in Brain Injured Patients
Acronym: NEGLECTARM3D
Status: Not yet recruiting | Type: Observational
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Other Study IDs: NEGLECTARM3D; PNC00000007 (Other Grant/Funding Number: Italian Ministry of University and Research)
Record Dates: First submitted 2025-11-21; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-09

CONDITIONS: Neglect; Brain Injured Patients; Stroke; Unilateral Spatial Neglect (USN); Post-stroke Cognitive Impairment
Keywords: Neglect; Brain injured patients; Tridimensional robotic assessment; Force-sensitive robot system; Virtual reality (VR) headset; Collaborative robotic system
MeSH Terms: conditions — Stroke | interventions — Physical Examination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- USN Patients Cohort: This single cohort includes patients diagnosed with Unilateral Spatial Neglect (USN) who are undergoing conventional neuromotor rehabilitation. The study involves the evaluation of a non-CE-marked robotic device to assess its usability and safety for three-dimensional assessment of USN, as well as to collect preliminary data on the reliability and validity of the device's measurements.
  Interventions: Device: Evaluation with a Non-CE-Marked Robotic Device

INTERVENTIONS:
Device: Evaluation with a Non-CE-Marked Robotic Device — Participants are assessed using a non-CE-marked robotic device to evaluate its usability and safety for three-dimensional assessment of Unilateral Spatial Neglect (USN), and to collect preliminary data on reliability and validity. This evaluation is part of the study and does not constitute an assigned intervention.

SUMMARY:
The goal of this clinical trial is to assess the usability and feasibility of a robotic and virtual reality-based system called NeglectARm 3D for the three-dimensional assessment of unilateral spatial neglect (USN) in patients with brain injury due to ischemic or hemorrhagic stroke.

The main questions it aims to answer are:

* Is the NeglectARm 3D system usable and feasible for patients with USN?
* Do the robotic measurements show preliminary reliability and validity compared with conventional clinical neglect assessments (e.g., BIT, CBS)?

Participants will:

* Perform two assessment sessions, three weeks apart (T0 and T1);
* Interact with the NeglectARm 3D system using a robotic end-effector and a VR headset to reach sequentially presented targets in a 3D virtual space;
* Receive robotic assistance if targets are not reached, allowing the system to record trajectories, spatial positions, and assistance applied;
* Complete standard clinical neglect tests to enable comparison between robotic and conventional measures.

This study aims to develop a repeatable, standardized, and objective tool for the assessment of USN in patients with brain injury, potentially improving evaluation of depth perception and spatial attention deficits.

DETAILED DESCRIPTION:
This observational, non-commercial study evaluates the usability and feasibility of the NeglectARm 3D system, a robotic and virtual reality-based tool for three-dimensional assessment of Unilateral Spatial Neglect (USN) in patients with brain injury due to ischemic or hemorrhagic stroke. Participants undergo two assessment sessions (T0 and T1), spaced three weeks apart, which include clinical neglect assessments using standard instruments and robotic evaluations with two test-retest trials per session.

The robotic component is the Franka Research 3 arm, a force-sensitive manipulator with seven degrees of freedom and torque sensors in each joint, providing industrial-quality pose repeatability of ±0.1 mm and minimal path deviation at high speeds. The virtual reality component is the Meta Quest 3 headset, which delivers high-resolution, smooth, and immersive visual feedback and tracks hand movement in real time using integrated sensors and RGB cameras.

During each session, participants reach sequentially presented stimuli in a 3D virtual space using their unaffected hand, in contact with the robotic end-effector. The system measures three-dimensional kinematics and provides assistance if the participant cannot reach a target independently. The robot operates in shared control mode, remaining transparent when the participant can reach a target autonomously ("patient-guided") and guiding the participant along the optimal trajectory when assistance is required ("robot-guided"), ensuring safe and natural movement.

The system records spatial positions and assistance parameters, enabling the construction of a map of target interactions and extraction of parameters for instrumental assessment of USN. Between assessment sessions, participants continue conventional rehabilitation. Data management includes checks for consistency and range, with source data verification performed by comparing robotic measurements with recorded observations. The study plans to enroll 15 patients, each completing two assessment sessions, to evaluate usability, feasibility, and preliminary reliability and validity of the system.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years;
* Diagnosis of ischemic or hemorrhagic stroke;
* Diagnosis of Unilateral Spatial Neglect (assessed by The Hearts Test, Oxford Cognitive Screen, cut-off ± 2);
* Signed informed consent form.

Exclusion Criteria:

* Presence of language deficits (inability to complete the OCS test);
* Presence of cognitive decline prior to the stroke event;
* Presence of severe visual and/or hearing impairments;
* Language barriers;
* Orthopedic, neurological, or psychiatric conditions that could interfere with the study or with the assessment of motor and cognitive function;
* Uncontrolled epilepsy despite antiepileptic treatment;
* Behavioral disorders that may interfere with study participation;
* Presence of medical devices whose functioning could be compromised (e.g., pacemaker, etc.);
* Object-centered neglect (assessed by the OCS Hearts Test; object asymmetry ± 2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The enrollment phase will be conducted at the IRCCS Fondazione Don Carlo Gnocchi in Florence (FI) and at the Fondazione Don Carlo Gnocchi in Sant'Angelo dei Lombardi (AV), in Italy. Each patient will be considered enrolled after assessment of inclusion and exclusion criteria and after signing the informed consent form. A total of 15 patients will be recruited, with 10 participants at the Florence center and 5 participants at the Sant'Angelo dei Lombardi center.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Usability of the NeglectARm 3D system | Baseline and 3 weeks from baseline
  Evaluation of usability of the NeglectARm 3D system using the HUBBI scale. The HUBBI (eHealth Usability Benchmarking Instrument) is a specialized tool for assessing the usability of eHealth services. It consists of 18 items rated on a 5-point Likert scale across seven key usability categories, focusing on the unique aspects of digital health platforms. This measure provides an indication of how repeatable, standardized, and safe the system is for the three-dimensional assessment of Unilateral Spatial Neglect (USN).
Feasibility of the NeglectARm 3D system | Baseline and 3 weeks from baseline
  Evaluation of feasibility of the NeglectARm 3D system, assessed by recording the type and number of side effects or system failures occurring during robotic evaluation. This measure provides an indication of how repeatable, standardized, and safe the system is for the three-dimensional assessment of Unilateral Spatial Neglect (USN).

SECONDARY OUTCOMES:
Behavioral Inattention Test (BIT) - Conventional subtest | Baseline and 3 weeks from baseline
  The BIT is a short screening battery of tests used to identify and quantify Unilateral Spatial Neglect (USN), consisting of 6 conventional paper-and-pencil subtests and 9 behavioral subtests.The BIT Conventional subtest consists of 6 items: line crossing, letter cancelation, star cancellation, figure and shape copying, line bisection, and representational drawing. It provides a maximum score of 146.
Catherine Bergego Scale (CBS) | Baseline and 3 weeks from baseline
  The Catherine Bergego Scale (CBS) is an observational tool designed to assess Unilateral Spatial Neglect (USN) in ecological contexts, such as activities of daily living. It consists of 10 items rated from 0 (no neglect) to 3 (severe neglect), with a maximum total score of 30; higher scores indicate greater neglect.
Motricity Index (MI) | Baseline and 3 weeks from baseline
  The Motricity Index (MI) is an ordinal method of measuring limb strength. For the upper extremity, shoulder abduction, elbow flexion, and pinch grip are considered; for the lower extremity, hip flexion, knee extension, and ankle dorsiflexion are considered. It ranges from 0 (worse) to 100 (normal strength). Measurements are taken bilaterally.
Montreal Cognitive Assessment (MoCA) | Baseline and 3 weeks from baseline
  The Montreal Cognitive Assessment (MoCA) is a widely used screening assessment for detecting cognitive impairment. It ranges from 0 (worst) to 30 (best).
Convergent validity between NeglectARm 3D measures and Behavioral Inattention Test (BIT) - Conventional subtest | Baseline and 3 weeks from baseline
  Convergent validity will be assessed by calculating correlation coefficients between instrumental (robot-based) measures of Unilateral Spatial Neglect (USN) recorded by the NeglectARm 3D system and the total score of the BIT Conventional subtest (BIT-C). Correlations between instrumental and clinical measures will be calculated using Pearson or Spearman correlation coefficients, depending on variable distribution. The outcome measure is the correlation coefficient between each instrumental measure and the BIT-C total score at each time point.
Convergent validity between NeglectARm 3D measures and Catherine Bergego Scale (CBS) | Baseline and 3 weeks from baseline
  Convergent validity will be assessed by calculating correlation coefficients between instrumental (robot-based) measures of Unilateral Spatial Neglect (USN) recorded by the NeglectARm 3D system and the total score of the CBS. Correlations between instrumental and clinical measures will be calculated using Pearson or Spearman correlation coefficients, depending on variable distribution. The outcome measure is the correlation coefficient between each instrumental measure and the CBS total score at each time point.
Test-retest reliability of total test execution time recorded by NeglectARm 3D | Within-session at baseline and within-session at 3 weeks from baseline
  Test-retest reliability of total test execution time recorded by the NeglectARm 3D system will be evaluated by comparing two repetitions of the robotic assessment performed within the same session at T0 and at T1. The outcome measure is the Intraclass Correlation Coefficient (ICC) between the two repetitions at each time point.
Test-retest reliability of number of targets identified without robotic assistance | Within-session at baseline and within-session at 3 weeks from baseline
  Test-retest reliability of the number of targets identified without robotic assistance during the NeglectARm 3D task will be evaluated by comparing two repetitions of the robotic assessment performed within the same session at T0 and at T1. The outcome measure is the Intraclass Correlation Coefficient (ICC) between the two repetitions at each time point.
Test-retest reliability of the number of targets not identified autonomously | Within-session at baseline and within-session at 3 weeks from baseline
  Test-retest reliability of the number of targets not identified autonomously (i.e., targets for which the robot had to provide assistance) during the NeglectARm 3D task will be evaluated by comparing two repetitions of the robotic assessment performed within the same session at T0 and at T1. The outcome measure is the Intraclass Correlation Coefficient (ICC) between the two repetitions at each time point.
Test-retest reliability of total robot intervention time | Within-session at baseline and within-session at 3 weeks from baseline
  Test-retest reliability of total robot intervention time during the NeglectARm 3D task will be evaluated by comparing two repetitions of the robotic assessment performed within the same session at T0 and at T1. The outcome measure is the Intraclass Correlation Coefficient (ICC) between the two repetitions at each time point.

CONTACTS AND LOCATIONS:
Overall Officials: Eugenio Falotico, PhD, Study Chair — Scuola Superiore Sant'Anna di Pisa
Locations (3):
- Italy (3):
  - Fondazione Don Carlo Gnocchi, Polo Specialistico Riabilitativo, Sant'Angelo dei Lombardi, AV
  - IRCSS Fondazione Don Carlo Gnocchi, Florence, FI
  - Scuola Superiore Sant'Anna, Pisa, PI

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kim YM, Chun MH, Yun GJ, Song YJ, Young HE. The effect of virtual reality training on unilateral spatial neglect in stroke patients. Ann Rehabil Med. 2011 Jun;35(3):309-15. doi: 10.5535/arm.2011.35.3.309. Epub 2011 Jun 30. PMID 22506138
- [Background] Chen ZJ, Gu MH, He C, Xiong CH, Xu J, Huang XL. Robot-Assisted Arm Training in Stroke Individuals With Unilateral Spatial Neglect: A Pilot Study. Front Neurol. 2021 Jul 8;12:691444. doi: 10.3389/fneur.2021.691444. eCollection 2021. PMID 34305798
- [Background] Fordell H, Bodin K, Eklund A, Malm J. RehAtt - scanning training for neglect enhanced by multi-sensory stimulation in Virtual Reality. Top Stroke Rehabil. 2016 Jun;23(3):191-9. doi: 10.1080/10749357.2016.1138670. Epub 2016 Mar 8. PMID 27077985